CLINICAL TRIAL: NCT01011569
Title: Randomized Controlled Trial of Cage Versus Plate in One Level Cervical Disc Disease
Brief Title: Comparison of Cage Versus Plate in One Level Cervical Disc Disease
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, Professor, Seoul National University Hospital
Other Study IDs: CAP trial
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Cervical Disc Disease
Keywords: difference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cage: patient who underwent stand alone cage insertion after discectomy
- plate: patient who underwent plate fixation and autologous ilia bone graft after discectomy

SUMMARY:
There are largely 2 surgical methods for one-level cervical disc disease; cage only and plate/graft. Even there are many reports about the efficacy of either cage only or plate/graft, prospective comparative study is few. The object of the present study is to present design of prospective study and to demonstrate preliminary result.

DETAILED DESCRIPTION:
Prospective study was started from April 2004 after permission by our Institutional Review Board. Inclusion criteria were single cervical disc disease with radiculopathy/myelopathy. We excluded patients with severe spondylosis, multiple disc disease, overt instability, osteoporosis or previous cervical operation history. Operation method was randomized using the table of random sampling numbers. All operations were performed with standard anterior-medial approach. Two types of cages and 2 types of plates were used: cage, MC+ cage (LDR, Austin, Tx, USA) or Solis cage (Stryker, Kalamazoo, Michigan, USA); plate, Black stone (Orthofix, McKinney, Tx, USA) or Atlantis (Medtronic, Minneapolis, MN, USA). We checked neck disability index (NDI), neck visual analogue scale (VAS) and limb VAS before operation and 1/3/6/12/24/36 months after operation. Disc height ratio, cervical lordosis, bone fusion status and segmental lordosis at the index level were measured from X-rays and follow-up X-rays were obtained at before operation and 1/3/6/12/24/36 months after operation. The present prospective study was planned until 80 patients (cage n = 40, plate/graft n = 40) were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were single cervical disc disease with radiculopathy/myelopathy.

Exclusion Criteria:

* We excluded patients with severe spondylosis, multiple disc disease, overt instability, osteoporosis or previous cervical operation history.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who needs surgery due to cervical disc disease
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2004-04; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Disc height ratio, cervical lordosis, bone fusion and segmental lordosis at the index level | 1/3/6/12/24/36 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Chun Kee Chung, professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Result] Kim CH, Chung CK, Hahn S. Autologous iliac bone graft with anterior plating is advantageous over the stand-alone cage for segmental lordosis in single-level cervical disc disease. Neurosurgery. 2013 Feb;72(2):257-65; discussion 266. doi: 10.1227/NEU.0b013e31827b94d4. PMID 23149973
- [Derived] Lee SE, Chung CK, Kim CH. Difference in canal encroachment by the fusion mass between anterior cervical discectomy and fusion with bone autograft and anterior plating, and stand-alone cage. J Clin Neurosci. 2016 Jul;29:121-7. doi: 10.1016/j.jocn.2015.10.039. Epub 2016 May 24. PMID 27234609